CLINICAL TRIAL: NCT06247085
Title: A Phase 3, Parallel-Group Treatment, Blinded, Randomized, Placebo-Controlled Study To Assess The Efficacy And Safety Of Pegtibatinase Administered Subcutaneously In Addition To Standard Of Care In Participants With Classical Homocystinuria Due To Cystathionine Beta Synthase Deficiency (HARMONY)
Brief Title: A Study to Investigate Efficacy and Safety of Pegtibatinase Compared With Placebo in Participants ≥12 to ≤65 Years of Age With Classical Homocystinuria (HCU) Due to Cystathionine Beta Synthase Deficiency Receiving Standard of Care Treatment
Acronym: HARMONY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVTX-TVT058-301
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Homocystinuria
Keywords: HCU; cystathionine beta synthase deficiency; Classical Homocystinuria
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- pegtibatinase (Experimental)
  Interventions: Drug: Pegtibatinase
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pegtibatinase — Full Target Dose of pegtibatinase BIW
  Other Names: OT-058; TVT-058
  Arms: pegtibatinase
Other: Placebo — volume-matched saline SC BIW
  Arms: placebo

SUMMARY:
The purpose of this study is to measure efficacy and safety of pegtibatinase treatment compared with placebo in participants with classical HCU receiving standard of care who have not achieved tHcy target levels. Study details include:

* Total Study duration: up to 38 weeks
* Screening:

  * Initial Screening duration: up to 4 weeks
  * Pre-treatment Diet Standardization Period duration: up to 6 weeks
* Blinded Treatment Duration: 24 weeks

  * 2-week blinded dose titration period
  * 22-week blinded assessment period
* Safety Follow-Up: 4 weeks after last dose (as applicable for those not enrolling in the long term extension study, ENSEMBLE)

DETAILED DESCRIPTION:
Overall Design:

This global Phase 3 multi-center, multi-national, randomized, blinded, placebo-controlled study will be conducted in participants with classical CBS deficient HCU receiving standard of care who continue to have tHcy levels ≥50 μM. The total study duration will be up to 38 weeks. Approximately 70 participants (35 per arm) will be randomized to receive active drug or placebo (1:1 allocation).

Screening:

Participants will enter into a 2-phase Screening period of up to 10 weeks:

1. Initial Screening: up to 4-week period during which participants will be assessed for eligibility
2. Pre-treatment Diet Standardization Period (DSP): After meeting initial eligibility criteria, participants will begin a pre treatment DSP of up to 6 weeks. The DSP is intended to help minimize variability in protein intake and supplements throughout the randomized portion of the study.

The baseline diet and compliance with HCU-related treatments will be recorded by the dietitian using the HCU-specific diet monitoring tool, called SING (Simplified Ingested Nutrients Guide). The baseline diet and treatment compliance will be used as a reference for future evaluation of daily intact protein intake (DIPI) and HCU treatments.

Blinded Treatment Period:

During the 24-week blinded treatment period, study visits will occur at regular intervals including home visits for study drug administration. Some study visits may be conducted remotely. Dietary protein intake and compliance with HCU treatments will continue to be monitored and recorded to ensure a stable diet and HCU treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥12 to ≤65 years of age, at the time of signing the informed consent
* Must have a diagnosis of classical HCU based on clinical, biochemical, and/or molecular genetic testing
* Plasma tHcy ≥80 µM at Screening visit, with allowance for up to 18 participants who may be enrolled with a Screening plasma tHcy ≥50 to <80 µM
* Willing to maintain a generally stable diet for the duration of the study (unless changes are required based on medical/safety reasons)
* Willing to maintain generally stable intake and doses of betaine, pyridoxine, and Met free formula for the duration of the study (unless changes are required based on medical/safety reasons)

Exclusion Criteria:

* Diagnosis of Marfan syndrome, methylenetetrahydrofolate reductase (MTHFR) deficiency, or disorder of cobalamin metabolism
* Concurrent disease or condition (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease) that would interfere with study participation or safety (excluding complications of HCU).
* History of major thrombotic event (eg, cerebrovascular accident, myocardial infarction, pulmonary embolism) in the previous 6 months.
* Body weight ≥160 kg.
* Use or planned use of any injectable drugs containing PEG (excluding PEG-containing vaccines)
* Any previous exposure to pegtibatinase and/or previous participation in a clinical study that included administration of pegtibatinase or pegtarviliase
* Prior severe immune reaction to a PEG-containing product

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plasma tHcy levels | Weeks 6 - 12
  The change from baseline in plasma tHcy levels averaged over Weeks 6 through 12 in participants receiving standard of care and treated with pegtibatinase as compared to participants receiving standard of care and placebo

SECONDARY OUTCOMES:
Plasma tHcy levels | Weeks 16 - 24
  The change from baseline in plasma tHcy levels averaged post Week 12 (Weeks 16, 20, 24)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Imperiale, MD, Study Director — Travere Therapeutics, Inc.
Locations (1):
- Travere Investigational Site - Virtual Site, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.